CLINICAL TRIAL: NCT05577052
Title: SBRT Versus Conventional Fractionated Radiotherapy for Vertebral Metastases From Non-small Cell Lung Cancer, an Open, Randomized Phase II Study
Brief Title: SBRT Versus Conventional Fractionated Radiotherapy for Vertebral Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Conghua Xie,MD,PhD, Professor, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBRT for vertebral metastases
Record Dates: First submitted 2022-10-08; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: NSCLC
Keywords: SBRT, NSCLC, Vertebral metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Metastatic vertebrae treated with SBRT
  Interventions: Radiation: Metastatic vertebrae treated with SBRT
- Control group (Other): Conventional radiation dose to vertebral metastases
  Interventions: Radiation: Metastatic vertebrae treated with SBRT

INTERVENTIONS:
Radiation: Metastatic vertebrae treated with SBRT — High-dose SBRT treatment

SUMMARY:
Vertebral metastases are events that affect the quality of life of tumor patients, and are often accompanied by severe pain at the site of metastasis and even by the risk of compression fracture. For vertebral metastases who are not yet at risk of vertebral instability fracture, a moderate dose (30Gy/10F) external radiation therapy is the most widely used treatment technique. Previous studies have shown that 60-80% of patients could achieve pain relief with moderate doses of radiation therapy, with median pain control duration of approximately 4 months. Stereotactic Radiation Therapy (SBRT) is currently the most advanced radiation therapy technique. This project proposes to treat vertebral metastases from non-small cell lung cancer using SBRT technology on the True Beam radiotherapy system to compare its efficacy with conventional external irradiation technology in terms of pain relief as well as local control.

DETAILED DESCRIPTION:
Vertebral metastases are events that affect the quality of life of tumor patients, and are often accompanied by severe pain at the site of metastasis and even by the risk of compression fracture. For vertebral metastases who are not yet at risk of vertebral instability fracture, a moderate dose (30Gy/10F) external radiation therapy is the most widely used treatment technique. Previous studies have shown that 60-80% of patients could achieve pain relief with moderate doses of radiation therapy, with median pain control duration of approximately 4 months.

Stereotactic Radiation Therapy (SBRT) is currently the most advanced radiation therapy technique. It enables focused radiation therapy with small fields through stereotactic techniques. In June 2021, Zhongnan Hospital of Wuhan University introduced the True Beam radiotherapy system, which has a higher treatment rate compared to conventional radiotherapy equipment, while It is the most reliable vehicle to achieve SBRT.

Therefore, this project proposes to treat vertebral metastases from non-small cell lung cancer using SBRT technology on the True Beam radiotherapy system to compare its efficacy with conventional external irradiation technology in terms of pain relief as well as local control.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed stage IV non-small cell lung cancer.
* General condition score ≤ 2.
* With vertebral metastases combined with painful symptoms.
* Absence of neurological symptoms due to vertebral metastases, such as dyskinesia, defecation or urination abnormalities.
* No previous radiation treatment of any kind to the vertebral body.
* The metastatic vertebra has not been treated surgically
* Vertebral stability score (SINS) ≤ 12
* Patient life expectancy of more than 6 months.

Exclusion Criteria:

* Small cell cell lung cancer or large cell carcinoma
* General condition score >2, intolerant of radiotherapy.
* Comorbid neurological symptoms such as dyskinesia, abnormal bowel movements or urination
* Metastatic vertebrae that have received radiotherapy or surgical intervention
* Vertebral stability score (SINS) >12
* Patient life expectancy of less than 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete pain relief rate | 3 months
  Complete pain relief rate after completion of radiotherapy

SECONDARY OUTCOMES:
Quality of life scores | 3 months and 6 months
  Quality of life score after radiotherapy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2 years of sharing after 3 months